**Study Title:** Identifying and addressing critical social, ethical, and behavioral factors associated with COVID-19 testing and vaccination among Spanish speakers

Principal Investigators: Scott D. Rhodes, PhD, MPH; Amanda E. Tanner, PhD, MPH

Co-investigators: Alain Bertoni, MD, MPH; Mark Hall, JD; Thomas P. McCoy, PhD

Sponsor or funding source: NIH

# **Background, Rationale and Context**

# Significance

Latinx communities in the US are disproportionately affected by COVID-19.5-7,33 Latinx (a gender-inclusive term34,35 that we use to refer to Hispanic/Latino populations in the US) persons comprise 18.5% of the US population and as of June 19, 2021, comprised 28.8% of US COVID-19 cases.36 Latinx persons are 2 times more likely to contract COVID-19 than their non-Latinx White counterparts, 2.8 times more likely to be hospitalized from COVID-19, and 2.3 times more likely to die from COVID-19.1 These disparities are even more profound among Spanish speakers and Spanish-speaking immigrants.1-7

Ongoing testing and vaccination are critical to effective control of the pandemic; however, complex issues contribute to low rates of COVID-19 testing and vaccination within Spanish-speaking Latinx communities.5-8,37 Factors that pose challenges to testing and vaccination include poverty, limited resources, and institutional and structural barriers (e.g., discrimination and limited transportation). Latinx persons may: lack access to culturally congruent information about COVID-19 testing and vaccination, including eligibility and how to access these services; believe they are not at risk for COVID-19; worry about missing work due to a positive test result or vaccine side-effects; and assume that they have to pay for a test or vaccine. Other challenges include fear of engaging with government systems (including public health) and of the long-term health implications of testing and vaccination. These barriers are even greater among those who do not speak English, are undocumented, and/or live in mixed-immigration status households.2,5-7,37 Our community-based participatory research (CBPR) partnership's preliminary research identified additional barriers, including: misinformation about testing and vaccination communicated through Spanish-language TV and social media and within social networks by word-of-mouth, and distrust in the test or vaccine (e.g., not believing that they will get the real vaccine as has happened in Latin America38,39; published2,40 and unpublished data).

A profound need remains to understand the social, ethical, and behavioral implications (SEBI) of COVID-19 testing and vaccination interventions within Spanish-speaking Latinx communities, 2.5,7,33,41-43 COVID-19 testing and vaccination are strongly influenced by social, ethical, and

**communities.**2,5,7,33,41-43 COVID-19 testing and vaccination are strongly influenced by social, ethical, and behavioral factors at the individual, interpersonal, institutional, community, and policy levels.44 While some of these multilevel factors are beginning to be explored, there is a great need for further empirical studies that focus on Spanish-speaking Latinx communities. The heterogeneity of the Latinx population is well established,34,35,45,46 and Spanish speakers experience markedly different barriers from other Latinx persons due to a range of factors such as more pronounced economic challenges, lower levels of acculturation, and heightened fear and mistrust of government systems (including public health). Furthermore, Spanish-speaking Latinx persons in the US may be undocumented and/or live in mixed immigration-status households35,47,48 and thus face unique challenges to testing and vaccination.

Peer navigation has potential to increase COVID-19 testing and vaccination within Latinx communities. Natural helping (e.g., peer navigation and lay health advising) is potentially effective in addressing health issues in underserved and vulnerable communities. 11,15,16,24,27,28,49-62 Peer navigation

harnesses relationships and networks to help individuals engage with prevention or care services. Peer navigators have advantages over other strategies because they can reach those who are considered "hard-to-reach" with carefully personalized messaging and support. As trusted community members, peer navigators can be the first people turned to for assistance. Effective peer navigators are part of the networks in which they work, in terms of self-identity, socioeconomic status, and lived experience; understand community needs and strengths and what is meaningful to members and communities; communicate in the language of members; and incorporate culture to promote positive behaviors.12,15,16,21,24,28,51,53,59,60,62,63 As our partnership has learned, peer navigation strategies can be sustainable, as peer navigators often continue their work after a study and funding end.23,64

mHealth can also be a powerful tool to reach Spanish speakers. Spanish speakers have high rates of social media use, including Facebook, Instagram, and texting, for acquiring health information,46,65-72 and this use extends to COVID-related information.2,42,73,74 These rates are related to increased proliferation of mobile devices, including among Spanish-speaking Latinx persons.75-77 Mobile devices support apps, including Facebook, which is the most commonly used social media platform.78 Because of its ubiquity and frequency of use, Facebook holds promise as a platform for health promotion.9,79-83 Facebook also has a direct messaging feature that allows users to communicate one-on-one and to a group. Instagram has also grown its user base and features. In addition to supporting photo and video sharing, Instagram offers a direct messaging feature, and Spanish speakers in our research recommend that we use this app in intervention implementation.12,70 At the same time, texting (including through messaging apps such as WhatsApp) continues to increase dramatically in all age groups and can be a powerful health promotion tool because it is widely available, inexpensive, and instantaneous, and can be effective at promoting behavior change.10,84-89

Because the health-related views of Latinx persons are strongly influenced by trusted social network members42,73,90 and because Spanish speakers are active users of social media, combining peer navigation with mHealth holds particular promise for increasing COVID-19 testing and vaccination within Spanish-speaking Latinx communities. Moreover, studies suggest that Latinx persons report increased willingness to be tested and vaccinated,91,92 indicating that focused support that addresses barriers and builds on facilitators could be highly effective. For example, in a recent national survey, eagerness to receive vaccination was more pronounced for Spanish-speaking Latinx persons than English-speaking Latinx persons (27% vs. 11%), but Spanish speakers reported greater information gaps and uncertainty about how orwhere to seek vaccination.92

This research is **significant** because Spanish-speaking Latinx communities carry disproportionate burdens of COVID-19 and have lower rates of testing and vaccination. However, there is limited understanding of the SEBI of testing and vaccination, and thus, a dearth of effective interventions to increase testing and vaccination within this population. Our study will fill these gaps through a better understanding of the individual, interpersonal, institutional, community, and policy factors influencing testing and vaccination and the testing of a Spanish-language intervention, known as *NuestraSaludSegura* (*Our Safe Health*), that integrates peer navigation and mHealth to increase testing and vaccination.

# Innovation

This study is innovative in several ways:

- 1) We focus on a distinctly underserved and vulnerable population the Spanish-speaking Latinx population who encounter multilevel barriers to COVID-19 testing and vaccination in the US.
- 2) This study is proposed by a well-established partnership that has been exploring multilevel factors influencing health and developing and testing interventions designed to promote health equity within Spanish-speaking Latinx communities using authentic CBPR for two decades.15,16,18,19,21,24,26,62,93-104
- 3) Our community partners and collaborators cover the entirety of NC, allowing us to capture a wide range of experiences and settings (e.g., urban, rural, and suburban) and increasing generalizability.

- 4) This study collects formative research designed to increase our understanding of the SEBI of COVID-19 testing and vaccination and immediately translates this understanding to *NuestraSaludSegura*, a novel intervention designed to increase testing and vaccination within Spanish-speaking Latinx communities.
- 5) The *NuestraSaludSegura* intervention harnesses the complementary strengths of peer navigation and mHealth to increase COVID-19 testing and vaccination. The underlying evidence for these strategies is emerging, and to our knowledge, they have not been applied in combination within general Spanish-speaking communities.
- 6) The intervention leverages social media via existing platforms that Spanish-speaking Latinx persons already use (e.g., Facebook, Instagram, and texting). Thus, the behavior change focuses on testing and vaccination behaviors, not the antecedent behavior of downloading, learning, and using a new "app", which some mHealth strategies rely on for implementation.
- 7) We also include a novel strategy to dissemination that our partnership has developed. Designed to be low burden for attendees, our theory-based community forum brings together community members, partners, and other stakeholders to review study findings and develop next steps for practice and research.95,100,105

# **Approach**

CBPR. CBPR has been identified as a critical approach to increase health equity and reduce disparities among underserved and vulnerable populations.16,26,94,103,104,106-118 Blending the lived experiences of community members, the expertise of service providers and public health practitioners, and sound science can develop deeper and more informed understandings of health and yield interventions that are more relevant, more culturally congruent, and more likely to be effective and sustained, if warranted.10,15,16,26,93,94,118-126 Furthermore, recruitment and retention rates may be higher, measurement may be more precise, data collection may be more acceptable, data analysis and interpretation of findings may be more accurate, and dissemination may be more likely than when using approaches that do not blend these multiple perspectives.94,111,117-119,126-129

The partners proposing this study have worked together for >18 years and have had many successes that, in part, we attribute to CBPR.26,96,103 We have engaged in intensive decision-making about all aspects of this study, including the qualitative methods (i.e., in-depth interviews and focus groups), the intervention strategies (i.e., peer navigation and mHealth) and evaluation methods (i.e., the longitudinal group-randomized trial design), and dissemination plans. We will continue to use CBPR throughout this study. Our partnership is not study-specific; members join and leave, and be more or less involved, but the partnership remains.10,11,26,96,100

The proposed study. We have created a conceptually integrated CBPR study that includes systematic data collection on the multilevel factors that influence COVID-19 testing and vaccination; refinement of an efficacious intervention that uses complementary theory-based strategies (i.e., peer navigation and mHealth); intervention implementation and evaluation using a longitudinal group-randomized trial design; and dissemination of findings. This is an ambitious study, and we have allocated sufficient effort and delineated clear roles and responsibilities among study team members and community partners to ensure we accomplish the Aims. As a community member noted, "We can't wait. COVID is hurting our community right now! We must do things that change these trends now!"

Catchment area. We will conduct this study across NC. NC has more than 1 million Latinx persons, many of whom are immigrants,139 and the COVID-19 experiences of its Latinx population reflect experiences nationally, increasing study generalizability.140,141 In NC, compared to other racial/ethnic groups, the rate of COVID-19 infections has been higher within the Latinx community and fewer Latinx persons have been vaccinated.142

Study-specific steering committee. This study will be guided by a study-specific steering committee. This committee will be comprised of representatives from the Latinx community, community-based organizations, and academic research institutions. We expect to have ~15 committee members. Our team has much expertise with facilitating study-specific steering committees.26,103,143 The committee will meet monthly to provide guidance on measurement; recruitment and retention; intervention refinement; and interpretation of findings. We will continue to use the "70%-consensus rule" to encourage consensus decision-making by asking if each committee member can support a decision by at least 70%.101,128

### **Objectives**

Aim 1: Collect, analyze, and interpret exploratory qualitative data to expand our understanding of the SEBI of COVID-19 testing and vaccination within Spanish-speaking Latinx communities. We will conduct 50 individual in-depth interviews with health providers (including administrators, clinicians, community health workers, and safety-net clinic staff) and with representatives from Latinx-serving community-based organizations; and conduct 6 focus groups with Spanish-speaking Latinx community members (total number of focus group participants=60).

Aim 2: Refine and test *NuestraSaludSegura* to determine its impact on COVID-19 testing and vaccination among Spanish-speaking Latinx persons using a group-randomized trial design.

Integrating our successes with peer navigation and mHealth strategies with other relevant COVID-19 studies and Aim 1 findings, we will refine and test the *NuestraSaludSegura* intervention. We will enroll 20 peer navigators, known as *Navegantes*, who represent 20 unique social networks, and 8 unique members from each social network for a total of n=160 social network members. After baseline data collection, we will randomize *Navegantes*, coupled with their social networks, into intervention and delayed-intervention groups (10 *Navegantes*; 80 social network members per group). We will train and support intervention-group *Navegantes* to increase COVID-19 testing and vaccination services within their social networks. We will evaluate the intervention by comparing changes in testing and vaccination from baseline to post-intervention follow-up between groups. *We hypothesize that intervention group will demonstrate increased COVID-19 testing and vaccination*.

Aim 3: Develop and disseminate practice, research, intervention, and policy priorities and recommendations to increase COVID-19 testing and vaccination among Spanish-speaking Latinx communities in the US. We will conduct an empowerment theory-based forum with Latinx community members and other community members and representatives from community-based organizations and universities to develop and disseminate priorities and recommendations based on study findings.

# **Methods and Measures**

### Design

### Aim 1:

We will conduct **individual in-depth interviews** with two categories of participants from across NC: (1) Health providers (including administrators, clinicians, community health workers, and safety-net clinic staff), who have planned, managed, and/or conducted COVID-19 testing and/or vaccination activities for Spanish-speaking communities; and (2) Representatives from Latinx-serving community-based organizations. We also will conduct **focus groups** with Spanish-speaking Latinx community participants.

### Aim 2:

We will refine and test the *NuestraSaludSegura* intervention, integrating our previous successes with peer navigation and mHealth strategies with other relevant COVID-19 studies and Aim 1 findings. We will then recruit, enroll, and collect baseline data from 20 *Navegantes* (peer navigators) and their social network members (n=8 unique social network members per *Navegante*) from across NC. *Navegantes* (coupled with their social networks) will be randomly assigned to: intervention or delayed-intervention groups (10 *Navegantes*; 80 social network members per group). Intervention-group *Navegantes* will be trained and supported for 6 months of implementation in Years 1-2; delayed-intervention group *Navegantes* will be trained in Year 2. CBPR partners emphasized that a delayed-intervention comparison design is the most equitable, acceptable, and ethical.

**Assessment of intervention efficacy.** We will use a longitudinal group-randomized trial design with 2 arms (intervention and delayed-intervention) to evaluate the impact of the intervention. Quantitative outcome data will be collected from each *Navegante* and their 8 enrolled social network members at 2 time points: (1) baseline (*prior* to randomization and *Navegante* training) and (2) immediate post-intervention (6 months after the *Navegantes* in the intervention group are trained).

**In-depth interviews**. After post-intervention follow-up, we will conduct in-depth interviews with each *Navegante* in the intervention group (N=10) to explore and better understand their implementation of the intervention, their natural helping behaviors, and other lessons learned.

### **Aim 3:**

The translation of findings into action is a CBPR hallmark,16,26,30,93-95,97,99,100,105,111,129,137,143,190-193 and we have developed an empowerment theory-based100,169,194,195 and highly collaborative process to do just that.95,100,166 We will organize and conduct a bilingual community forum to translate findings into practice, research, intervention, and policy priorities and recommendations.

### **Setting**

The study will take place in community settings (e.g., community organizations) across NC.

### **Subjects selection criteria**

### • Inclusion Criteria

### Aim 1:

To be eligible to participate in the <u>in-depth interviews</u> as a health provider, a participant must (a) be employed at a clinic, health center, or other organization that has planned, managed, and/or conducted COVID-19 testing and/or vaccination activities for Spanish-speaking communities; (b) be  $\geq$ 18 years of age; and (c) be willing to participate. To be eligible to participate in the interviews as a Latinx-serving community-based organization representative, a participant must (a) be affiliated with a Latinx-serving community-based organization, (b) be  $\geq$  18 years of age, and (c) be willing to participate.

To be eligible to participate in the <u>focus groups</u>, a participant must (a) self-identify as Hispanic/Latinx, (b) be Spanish speaking, (c) be  $\ge 18$  years of age, and (d) provide informed consent.

### **Aim 2:**

To be eligible to participate in the *NuestraSaludSegura* intervention as a *Navegante*, a participant must (a) self-identify as Hispanic/Latinx, (b) be Spanish speaking, (c) be  $\geq 18$  years of age, (d) provide informed consent, and (e) report having been vaccinated against COVID-19 (because *Navegantes* serve as role models). Access to a smartphone will not be an inclusion criterion. We have some flexibility to provide smartphones and data plans for *Navegantes* without them, though given smartphone proliferation (and our past research experiences), this will likely be unnecessary.

To be eligible to participate in the intervention as a *social network member*, a participant must (a) self-identify as Hispanic/Latinx, (b) be Spanish speaking, (c) be  $\geq 18$  years of age, and (d) provide informed consent.

# • Sample Size

### Aim 1:

We will conduct **50 individual in-depth interviews** for a total number of 50 interview participants and **6 focus groups** with 8-12 participants each for a total number of 60 focus group participants. We will screen participants to ensure we obtain representation by: gender, documentation status, and those with and without experiences of COVID-19 testing and vaccination. As it is difficult to predict **saturation**<sub>144-150</sub> *a priori*, we have flexibility to expand the number of interviews and/or focus groups if warranted. Project members working with the qualitative data will meet regularly to discuss emerging themes and determine if saturation has been reached.

### **Aim 2:**

Sample size calculations are based on a follow-up adjusted baseline (or ANCOVA) model. We estimated the sample size needed (20 *Navegantes* and 160 social network members) by performing calculations in nQuery v8.7.

# **Interventions and Interactions**

# Aim 1:

Interviews will be digitally recorded. While interviews and focus groups can be conducted remotely via telephone and videoconferencing platforms (e.g., Zoom and WebEx), we will conduct them in-person if possible based on the current CDC recommendations. Safety precautions (e.g., personal protective equipment) will be followed as indicated. Dr. Rhodes and an infectious disease epidemiologist published guidelines for safely conducting community-based and community-engaged in-person research during COVID,151 which have been adopted by multiple Clinical and Translational Science Award hubs throughout the US and by CDC research teams.

The in-depth interview and focus groups guides. These guides will be structured to gather *descriptive* "deep"<sub>152</sub> qualitative data. An initial low-literacy assessment will collect demographic data. Guides will be developed iteratively with the steering committee and in consultation with the RADx-UP Coordination and Data Collection Center (CDCC) and consortium through ongoing literature review; brainstorming of domains and constructs; and drafting, review, and revision of potential questions. Because this Aim is

**exploratory** and designed to be **inductive**, the framework is subject to revision. This Aim's outcome will be a better understanding of the SEBI of COVID- 19 testing and vaccination among Spanish- speaking Latinx persons. Interview guides will adhere to best practices (e.g., creating non-leading/open-ended questions, ordering from general to specific, maintaining neutral tone, and depersonalizing behaviors by third-person-ing questions) to elicit knowledge, descriptions of experiences, opinions, and values.98.146.150.153-156

### Aim 2:

The original intervention and its refinement. The bilingual weCare intervention serves as a foundation for NuestraSaludSegura. weCare is based on the social cognitive and empowerment theories and social support9,10,28,168-170 and harnesses peer navigation and mHealth.9-14 The objectives of weCare (i.e., to increase care engagement and improve health outcomes among vulnerable persons with HIV) align with the objectives of NuestraSaludSegura (i.e., to increase testing and vaccination among vulnerable persons disproportionately impacted by COVID-19). Thus, the refinement process will be efficient and include revising the Navegante training and mHealth messages. The study team and the steering committee will conduct the refinement in parallel to Aim 1, integrating findings from other relevant studies(e.g., 69,171,172) and from Aim 1 as they emerge. Specifically, we will review the theoretical underpinnings of the intervention and anticipated outcomes of NuestraSaludSegura and refine the training, including the mHealth messages, to build Navegante capacity to increase COVID-19 testing and vaccination within their social networks. This process is designed to expedite the translation of Aim 1 findings into intervention, which is a hallmark of CBPR94,113 and a priority of our partnership given the burden of COVID-19 within Spanish-speaking Latinx communities.

Each *Navegante* will serve as a health advisor, opinion leader, and community advocate and use in-person and/or virtual (through Facetime or Zoom) individual and group activities and mHealth (using Facebook messenger, Instagram direct messaging, and text messaging) to communicate and provide social support within their social networks during the 6-month intervention. The *Navegantes* approach is personalized to each social network member's needs and priorities. **Table 1** provides an abbreviated summary of *Navegante* activities and examples of activities operationalized.

Based on our partnership's history training peer navigators,15-28 we currently have a *Navegante Training Manual*, which will guide the 4-session interactive training of the *Navegantes*, including sections on effective facilitation, how to prepare for training, session checklists, and all training activities and materials. This manual will require refinements related to COVID-19. We also will develop a *Navegante Resource Guide* that will provide details about COVID-19 testing and vaccination across NC (e.g., local providers and services and eligibility information) that *Navegantes* can refer to as they work with their social networks after training.

We will refine our *weCare* library of theory-based sample messages<sub>10</sub> that *Navegantes* can tailor and use to meet the specific needs of each social network member. We have much experience with mHealth message development to improve health outcomes.<sub>9,10,12,14,29,99,135,173</sub> A critical component of *NuestraSaludSegura* is the "connection" between the *Navegantes* and social network members. Growing evidence suggests that in-real-time, personalized, and bidirectional social support and problem solving provided by a peer using mHealth may be more successful in changing behaviors among populations facing many multilevel barriers to change than other technology-based approaches, such as software applications providing automated messages.<sub>12,14,29,174-176</sub> In our research to better understand the mechanisms underlying *weCare*, we discovered the importance of participants "knowing the person behind the messaging" and perceiving that this person cares about them.<sub>12</sub>

Table 1. Activities of Navegantes in the NuestraSaludSegura intervention

# Activities Raise awareness of the ongoing need for COVID-19 testing and vaccination Provide information and referrals De-mystify the process of seeking COVID-19 testing and vaccination Reframe and bolster norms and expectations

### Share announcements and reminders

Troubleshoot and problem solve SEBI of COVID-19 testing and vaccination

Support communication with providers and staff

Support other prevention behaviors

Provide feedback to providers and staff

### **Examples**

Navegantes increase consciousness among their social networks about the need for testing and vaccination to slow the spread of COVID-19, state and local rates of testing and vaccination and among Latinx populations, and the importance of taking action.

Navegantes provide information about local providers of COVID-19 testing and vaccination services (e.g., testing and vaccination sites near a social network member's home or workplace, days and hours of operation, and whether an appointment is needed and how to make one).

Navegantes explain what to expect when accessing COVID-19 testing and vaccination, including where to go, how to get there by public transportation (or where to park if in a car), the presence of security, sign-in processes, what information will be requested (e.g., if staff will ask for identification or insurance information), availability of interpreters or Spanish-speaking staff, what steps are involved in the testing or vaccination process, and how long the process will take (e.g., turnaround time for receiving test results and required observation period after receiving the vaccine).

Navegantes highlight how the benefits of COVID-19 testing and vaccination are linked to social network members' priorities (e.g., protecting the health of their families and communities and facilitating the ability to gather with others safely). Navegantes share announcements with social network members about upcoming testing and vaccination events. Navegantes help overcome stigma related to COVID-19 and build trust around testing and vaccination (e.g., addressing concerns about immigration status and confidentiality). Navegantes brainstorm options for overcoming barriers related to transportation (e.g., if a COVID-19 testing or vaccination site is not on a bus line and a social network member does not have a car or a driver's license), schedules (e.g., conflicts between work schedules and testing or vaccination site hours), and other challenges (e.g., concerns about the potential impact of a positive COVID-19 test result or vaccine side effects on the ability to work).

Navegantes talk through ways to effectively communicate and share concerns with providers and staff at testing and vaccination sites. Navegantes may remind social network members to bring a list of questions, symptoms, or information about potential COVID-19 exposures when going to get tested or vaccinated.

*Navegantes* provide guidance on recommendations for other prevention behaviors (aligning with current CDC guidelines), including mask use, social distancing, and potential need for booster vaccination.

Navegantes meet with providers and staff at COVID-19 testing and vaccination sites to provide feedback for multilevel changes to improve accessibility for Spanish-speaking Latinx communities.

**Baseline and immediate post-intervention assessment.** We will develop a Spanish-language assessment to collect data at baseline and immediate post-intervention (6 months post-baseline), based on Aim 1 findings, other relevant studies describing factors influencing COVID-19 testing and vaccination, our previous successes with peer navigation and mHealth strategies, and the theories underlying the intervention. **Table 2** outlines *draft* measurement priorities identified by our partnership while preparing this application. To ensure data harmonization, we will use the RADx-UP Common Data Elements and PhenX toolkit (https://www.phenxtoolkit.org/). The assessment, including final selection of measures,

Protocol version: Template updated 9.24.14 will be created using an *iterative* process by partners, including consultation with the RADx-UP CDCC and consortium

Table 2. Measurement priorities

Other variables

Outcome variables Primary: COVID-19 testing and vaccination including ever being tested, ever being vaccinated,

being up to date on recommended doses, and number of doses received

Demographic variables Age and date of birth; birthplace; ethnicity/race; language use; current living situation; zip code;

marital/partner status; family structure (e.g., children); educational attainment; current employment; financial status; immigration status; pregnancy status; insurance status

Symptoms COVID-19 symptoms and exposure to assess need for testing

Potentially mediating Awareness and knowledge about risk, testing, and prevention of COVID-19; intentions and variables readiness for COVID-19 testing and vaccination; perceived COVID-19 testing and vaccine a

readiness for COVID-19 testing and vaccination; perceived COVID-19 testing and vaccine access; knowledge of how to access testing and vaccination services; service use self-efficacy; perceived barriers to services; usual source of care; skills and self-efficacy to communicate effectively with providers; provider trust; history seeking and using prevention and care services; self-efficacy to overcome barriers; perceived provider discrimination; stigma related to COVID-19; social support; community attachment; perceived impact of positive test on job security; access to transportation

Intervention acceptability; satisfaction with participation in intervention; interactions with

Navegante and social network members regarding COVID-19 testing and vaccination (to assess

contamination)

Navegante training and support. The Navegante training will be designed to increase knowledge and build skills as health advisors, opinion leaders, and community advocates in person and/or virtually and through mHealth. Navegantes will be trained to use a version of the "ask-advise-assist" model to provide guidance and help others and will be given a wallet-sized reminder card that outlines the steps, as we have done within peer navigation interventions in the past.19,70 Trained Navegantes will then carry out helping activities to increase COVID-19 testing and vaccination within their social networks for 6 months. During this time, Navegantes will be supported and meet with study staff as a group (monthly) and individually (as needed) for social support, intervention planning, experience sharing, and problem solving in person, virtually, by phone, and/or by social media. As part of the process evaluation, they will submit monthly Activity Logs (described below) to document their work with members of their social networks.(e.g., 20,50)

How will the trained Navegantes increase COVID-19 testing and vaccination within social networks? Through informal individual interactions and more formal activities, Navegantes will fulfill multiple roles. First, as health advisors, Navegantes will raise social network members' awareness of the ongoing need for COVID-19 testing and vaccination and help them think through pros and cons and how to overcome commonly experienced barriers to accessing services. For example, a social network member may hesitate to seek testing because they fear disclosing their immigration status or do not trust providers. Thus, the *Navegante* will describe what is required for testing and how providers are required to maintain confidentiality. As opinion leaders, Navegantes will reframe and bolster norms and expectations about COVID-19, testing, and vaccination. Navegantes are taught the concept of reciprocal determinism from social cognitive theory 168 to illustrate how attitudes and behaviors are influenced by and influence one's environment. For example, some Spanish speakers may have fatalistic views about COVID-19; thus, a *Navegante* may reframe attitudes regarding COVID-19 to encourage testing and vaccination as taking control of one's health. Third, as community advocates, *Navegantes* will bring the voices of Spanish speakers to providers. Navegantes will participate in tours of local testing and vaccination site within their region, which will provide Navegantes direct experiences with accessing services that will help them support their social network members in using services, build relationships between Navegantes and providers, and provide opportunities for Navegantes to share feedback for process improvement (based on their own experiences, the experiences of their social network members, as well as Aim 1 findings) with providers over time.

Each *Navegante* will also conduct group activities in-person and/or virtually with their social network members including an initial meeting to "inaugurate" their role as a community resource. Study staff will

Protocol version: Template updated 9.24.14 provide guidance to the *Navegantes* and assist them in conducting group activities. These activities will be documented on the Activity Logs (described below) that will provide important details for intervention evaluation, especially because not every social network member will attend each session.

In addition to in-person and/or virtual individual and group activities, *Navegantes* will use the mHealth platform(s) preferred by each social network member (i.e., Facebook, Instagram, and/or texting) to communicate directly with them during the intervention to plan activities and support use of COVID-19 testing and vaccination services. For example, *Navegantes* will use social media to remind social network members about group activities and problem solve attendance challenges. A *Navegante* and social network member may also communicate "in-real-time" via social media about the process of receiving COVID-19 testing and vaccination; for example, the *Navegante* may help the social network member navigate a clinic. The *Navegantes*' ability to provide immediate, efficient, and bidirectional communication is critical to overcome barriers to taking action and initiating service use.

Each *Navegante* will also use personalized Facebook and Instagram accounts for indirect communication (e.g., posting information about COVID-19 testing and vaccination events). In our *weCare* intervention, we learned that study-specific Facebook pages are less effective than accounts that function like a personal Facebook profile. In addition to being low literacy, Facebook and Instagram posts will be engaging and informative. For example, graphics that illustrate the rates of COVID-19 testing and vaccination in different population subgroups can raise awareness of the importance of taking action. We will provide *Navegantes* with links to reliable sources, including CDC and state COVID-19 informational websites. *Navegantes* will also post informal and welcoming pictures and videos (recorded using smartphones) of local COVID-19 testing and vaccination services staff and facilities to demystify what it is like to access services and to increase self-efficacy to use services. While it is possible that not all participants use all social media platforms, given the current use of Facebook and Instagram, and their potential as low burden communication methods, these posts will be worthwhile. Furthermore, they may reach others who are not enrolled in this study. All posted information will be correct, consistent, and linked to the intervention's theoretical underpinnings; study staff will be available to help *Navegantes* think through their messaging.

Activity Logs. Navegantes will complete and submit monthly Activity Logs. Activity Logs aid in our process evaluation and serve as triggers for Navegantes to initiate activities. 20,50 They document whom the Navegante worked with for each activity (e.g., codes for those within and outside of the enrolled social network members); the type of helping activity; whether it was an individual or group activity (and the number of people involved); and whether, which, and how mHealth platforms were used. Importantly, the Activity Log will allow us to assess the Navegantes' work beyond their enrolled social network members. An innovation of this study is that we will be able to precisely describe what the Navegantes did and who was reached.

**In-depth interviews with** *Navegantes*. In-depth interview guide development and data collection with *Navegantes* will mirror the processes described above in Aim 1.

### **Aim 3:**

We will invite partnership members, organization representatives (e.g., providers and clinic and community organization staff), community members, and academic researchers, to review and discuss study findings. As a group, they will respond to 4 empowerment theory-based trigger questions that move from concrete ("What do you see in these findings?" "In what ways do these findings make/not make sense to you?") to action ("What can be done?" "What can we do?"). Based on the triggers, attendees will brainstorm specific strategies. Next, using a nominal group process,21,95,100,105,196 attendees will define practice, research, intervention, and policy priorities for next steps based on 2 criteria (*importance* and

feasibility) 95,100,197-199 to ensure priorities have potential to decrease COVID-19 disparities. Examples of priorities that may emerge include social marketing/social media campaigns; clinical staff training to reduce perceived discrimination, better assess risk, and/or problem solve particular testing and vaccination access challenges experienced by Spanish-speaking Latinx persons; development of culturally congruent COVID-19 educational materials; and additional interventions (e.g., to reduce stigma) to increase adherence to recommendations.

Attendees will then divide into small groups based on the identified priorities, develop recommendations for carrying out those priorities, and present plans to the larger group of attendees. Action plans may include a timeline for next steps or a list of other individuals and organizations to engage. The forum also may identify priorities for future research and intervention development.

# **Outcome Measure(s)**

Primary outcome measures are COVID-19 testing and vaccination, including ever being tested, ever being vaccinated, being up to date on recommended doses, and number of doses received.

# **Analytical Plan**

### **Aim 1:**

**In-depth interview and focus group data analysis.** We will analyze the qualitative data using constant comparison, a systematic approach to developing grounded theory<sub>144,157</sub> that is well-suited to uncovering participants' meanings and experiences. 144,157,158 It combines inductive coding with simultaneous comparison; initial observations are continually refined throughout data collection and analysis. 149,157,159 The goal is to identify themes, not to quantify participant experiences. 12,62,160,161 Analytical steps include:

- Interviewers will document post-interview and focus group impressions (e.g., content, process, and themes).
- Interviews and focus groups will be professionally transcribed and translated (if needed). Translation allows for simultaneous, collaborative analysis and iterative discussion of themes to yield more accurate findings.
- Interviewers will verify transcripts by reviewing and correcting discrepancies while listening to the recording.
- Transcripts will be managed using the NVivo (Chicago, IL) and examined to identify and code domains for theme development. 145,163 This will begin with analysts reading the same 3 transcripts and writing memos (written records of the analysis process linked to the specific transcript). These represent conceptual, theoretical, and operational notes to help compare domains within and across interviews and focus groups and inform the initial analytical coding scheme. 144
- The analysts will meet to develop a common coding system and data dictionary.
- All transcripts will be coded by at least 2 analysts (allowing for the addition of emerging codes).
- For data triangulation, analysts will develop, compare, then revise matrices that identify similarities and differences and explore emic and etic perspectives within and across participant categories (e.g., health providers v. Latinx-serving community-based organization representatives; health provider/organization representative interview v. Spanish-speaking Latinx community member focus group).160
- The CBPR partnership will review themes for validity (e.g., rigor, credibility, and trustworthiness).97,164-167

Aim 1 draws from a rich and thorough set of state-wide experiences that reflect millions of testing and vaccination encounters and the diverse perspectives of Spanish speakers and those who directly serve them across a wide range of settings. Thus, it will accomplish the most comprehensive qualitative assessment to date of SEBI of COVID-19 testing and vaccination among Spanish-speakers. Our results, in addition to informing Aim 2, will be important in their own right to inform other researchers and practitioners. Accordingly, results from Aim 1 will be shared as soon as available with RADx-UP CDCC and consortium.

### **Aim 2:**

**Hypotheses.** We anticipate that participants in the intervention group, relative to their counterparts in the delayed-intervention group, will demonstrate increased COVID-19 testing and vaccination.

**Quantitative data analysis plan.** Data analysis will include **study group description** and **intervention impact evaluation**. *Study group description*. Frequencies and percentages for categorical variables and means, medians, standard deviations, and ranges for continuous variables will be tabulated to describe the sample. Reliability for measures will be estimated via internal consistency using coefficients alpha and omega. 178 Baseline intervention and delayed-intervention group comparisons will be performed. Correlation analyses will evaluate the associations between pairs of variables. Nonparametric statistics will be used when appropriate to evaluate significance of associations.

Evaluation of intervention impact. Data will be analyzed with an intent-to-treat approach.179 Randomization at the social network level will likely balance cluster-level baseline characteristics; however, as randomization may not precisely balance these, and there may be differences in social network member characteristics after network randomization, inverse probability weighting using propensity scores will be explored to balance baseline characteristics (both network and individual) between arms<sub>180</sub> using best practices.<sub>181</sub> Balance on propensity scores between intervention groups will be assessed using standardized differences.182 Propensity scores have been used in cluster RCTs.183 We will evaluate the intervention impact by comparing rates of past 6-month COVID-19 testing and vaccination completion (defined as complete dosage of approved vaccination: e.g., 2 Pfizer or Moderna doses or 1 Johnson & Johnson dose) between intervention and delayed-intervention group social network members at immediate post intervention (6 months after the intervention group *Navegantes* are trained), adjusting for baseline rates. This ANCOVA approach has the advantage of being unaffected by baseline differences; if baseline rates, by chance, were different, the intervention effect would be overestimated by looking at change scores and underestimated by a follow-up score analysis. The ANCOVA approach gives the same answer regardless of baseline imbalance. Additionally, the approach generally has greater statistical power to detect an intervention effect than the other methods. 184 Statistical analysis will be performed using generalized linear mixed modeling 185 for binary outcomes (sometimes termed randomeffects logistic regression). These models can assume a logit link for binary data (i.e., tested or vaccinated in past 6 months: yes/no) and allow for accounting for the within-group association of outcomes. If participants have repeated COVID-19 testing performed then an additional random effect for multiple testing will be considered, where appropriate. The generalized linear mixed model is an extension of general linear models that allows for non-independence of observations (e.g., within social networks).

The hypothesis that intervention and delayed-intervention groups differ in their prevalence, p, of COVID-19 testing or vaccination will be tested with the mixed-effects logistic model: Logit  $(p_{ij}l) = \beta_0 + \beta_1 Y_{ijo} + \beta_2 INTVN + v_i$ , where  $p_{ij}l$  is the probability of testing or vaccination at immediate post-intervention for participant i in social network j,  $Y_{ij0}$  is 1 if participant i in social network j reports testing or vaccination at baseline and 0 otherwise, and, INTVN =1 for the intervention group and 0 for the delayed-intervention group. The random effect  $v_j$  is the random effect for participants in social network j. The variance component for this random effect addresses the within-social network correlation. Under this model,  $\beta_2$ 

corresponds to the difference in prevalence of testing or vaccination at immediate post-intervention between the intervention and delayed-intervention groups on the logit scale. This random-effects logistic regression model will be fit using adaptive Gaussian quadrature in SAS PROC GLIMMIX.186

This regression approach will allow us to produce estimates of prevalence and prevalence change additionally *adjusting for individual and cluster-level covariates*, which will be compared to unadjusted estimates. Individual-level covariates may include age, country of origin, employment status, and education level. Because there are only a small number of clusters (social networks), the literature advises that the number of cluster-level covariates should be limited to one or two key variables. 187, 188 To assess the importance of covariates, we will use a backwards elimination model building approach, with primary consideration on assessment of confounding on the intervention-group difference. If confounding is present (defined to be greater than a 10% change in the regression estimate of the intervention-group effect), the confounder will be retained in the multivariable model. If many confounders are retained, alternative/sensitivity analyses will be conducted using propensity score weighting. All analyses will be 2-sided. 189 Note: While a better understanding of the relationships between members of social networks can be interesting, social network analysis is beyond the scope of this proposal based on our hypotheses and analysis plans.

Quantitative data collection/management. Assessment data will be collected by the study team in a safe and private location using audio-computer-assisted self-interview (ACASI) technology. We most recently used ACASI in our *weCare* intervention for English and Spanish data collection<sub>9-14</sub> and have worked out logistical details (e.g., data saving and backup) and ways to maintain participant interest. ACASI data collection overcomes challenges of literacy and will be conducted in Spanish. Saved ACASI files will be transferred using the Warehouse Manager to SAS data files for analysis and stored on a password protected secure server.

**In-depth interview data analysis**. Analysis of the data from in-depth interviews with *Navegantes* will mirror the qualitative data analysis processes described above in Aim 1.

### **Aim 3:**

We will develop a final report of findings and practice, research, intervention, and policy priorities and recommendations to distribute to attendees, the RADx-UP CDCC and consortium, and others for whom the findings will be relevant (e.g., local and state-level health department leaders). We successfully used this approach previously to translate findings into action in a study of HIV disparities among sexual minority men. Subsequent actions led by forum attendees were (1) redirection of NC state prevention funds to develop safe spaces for facilitated group dialogue around intimacy and HIV risk; (2) a statewide conference to develop advocacy skills among community leaders; and (3) a new research partnership to explore the impact of immigration policy on healthcare use within Latinx communities.26,100

# **Human Subjects Protection**

# **Subject Recruitment Methods**

### Aim 1:

In-depth interview and focus group participants for Aim 1 will be recruited through our partnership's broad networks of collaborators and community partners and by word-of-mouth.

### **Aim 2:**

Protocol version: Template updated 9.24.14 Intervention participants for Aim 2 can be recruited as a *Navegante* or social network member of a *Navegante*. Potential *Navegantes* will be recruited by being invited to an individual interview in which we will explore eligibility and personal, performance, and situational characteristics relevant to serving as a *Navegante*. We will then select *Navegantes*. After enrolling, each *Navegante* will be provided a script and recruitment materials to present to their social network members, explaining the study and asking them to contact staff using the study's toll-free number to enroll.

# **Informed Consent**

Verbal informed consent will be obtained from each focus group participant, and signed informed consent will be obtained from each Navegante and each social network member participant. The investigators or other study staff will obtain informed consent in community-based settings before collecting data from participants.

Interview participants will be provided with a brief description of the study to review before deciding to participate.

# **Confidentiality and Privacy**

Confidentiality will be protected by collecting only information needed to assess study outcomes, minimizing to the fullest extent possible the collection of any information that could directly identify subjects, and maintaining all study information in a secure manner. To help ensure subject privacy and confidentiality, only a unique study identifier will appear on the data collection form. Any collected patient identifying information corresponding to the unique study identifier will be maintained on a linkage file, store separately from the data. The linkage file will be kept secure, with access limited to designated study personnel. Following data collection subject identifying information will be destroyed six years after closure of the study, consistent with data validation and study design, producing an anonymous analytical data set. Data access will be limited to study staff. Data and records will be kept locked and secured, with any computer data password protected. No reference to any individual participant will appear in reports, presentations, or publications that may arise from the study. A limited dataset will be sent to the CDCC via a secure web portal. Data will be stored by the CDCC on protected, secure computer systems. Anyone with permission to see these data will have to use a password and multi-factor authentication.

### **Data and Safety Monitoring**

The principal investigator will be responsible for the overall monitoring of the data and safety of study participants. The principal investigator will be assisted by other members of the study staff.

# Reporting of Unanticipated Problems, Adverse Events or Deviations

Any unanticipated problems, serious and unexpected adverse events, deviations or protocol changes will be promptly reported by the principal investigator or designated member of the research team to the IRB and sponsor or appropriate government agency if appropriate.

### References

- 1. National Center for Immunization and Respiratory Diseases C. *Risk for COVID-19 Infection, Hospitalization, and Death By Race/Ethnicity*. Atlanta, GA. 2021.
- 2. Rhodes SD, Mann-Jackson L, Alonzo J, Garcia M, Tanner AE, Smart BD, Horridge DN, Van Dam CN, Wilkin AM. A rapid qualitative assessment of the impact of the COVID-19 pandemic on a

- racially/ethnically diverse sample of gay, bisexual, and other men who have sex with men living with HIV in the US South. *AIDS Behav.* 2021;25(1):58-67.
- 3. Barry K, McCarthy M, Melikian G, Almeida-Monroe V, Leonard M, De Groot AS. Responding to COVID-19 in an uninsured Hispanic/Latino community: Testing, education and telehealth at a free clinic in Providence. *R I Med J.* 2020;103(9):41-46.
- 4. Mehring WM, Kim JS, Hendel C, Hochman M. COVID-19 exposure risk by speakers of Spanish and English using a web-based self-assessment tool. *J Gen Intern Med.* 2021;36(6):1835-1836.
- 5. Rodriguez-Diaz CE, Guilamo-Ramos V, Mena L, et al. Risk for COVID-19 infection and death among Latinos in the United States: Examining heterogeneity in transmission dynamics. *Ann Epidemiol*. 2020;52:46-53.e42.
- 6. Hamel L, Artiga S, Satarpour A, Stokes M, Brodie M. *KFF COVID-19 Vaccine Monitor: COVID-19 Vaccine Access, Information, and Experiences Among Hispanic Adults in the U.S.* San Francisco, CA: Kaiser Family Foundation. 2021.
- 7. Reitsma MB, Claypool AL, Vargo J, et al. Racial/ethnic disparities in COVID-19 exposure risk, testing, and cases at the subcounty level in California. *Health Aff.* 2021;40(6):870-878.
- 8. Oelsner EC, Allen NB, Ali T,... Bertoni AG, et al. Collaborative Cohort of Cohorts for COVID-19 Research (C4R) Study: Study design. *medRxiv*. 2021.
- 9. Tanner AE, Mann L, Song E, Alonzo J, Schafer K, Arellano E, Garcia M, Rhodes SD. weCare: A social media-based intervention designed to increase HIV care linkage, retention, and health outcomes for racially and ethnically diverse young MSM. *AIDS Educ Prev.* 2016;28(3):216-230.
- 10. Tanner AE, Song EY, Mann-Jackson L, Alonzo J, Schafer KR, Ware S, Garcia M, Arellano Hall E, Bell JC, Van Dam CN, Rhodes SD. Preliminary impact of the weCare social media intervention to support health for young men who have sex with men and transgender women with HIV. *AIDS Pt Care STDs.* 2018;32(11):450-458.
- 11. Alonzo J, Mann-Jackson L, Garcia M, Tanner AE, Rhodes SD. Atendiendo las necesidades de jóvenes latinos gay, bisexuales y otros hombres que tienen sexo con hombres (HSH) y mujeres transgénero que viven con VIH a través de la intervención weCare en los Estados Unidos (EEUU). *EHQUIDAD*. 2021;15:209-232.
- 12. Tanner AE, Mann-Jackson L, Song EY, Alonzo J, Schafer KR, Ware S, Horridge DN, Garcia JM, Bell J, Hall EA, Baker LS, Rhodes SD. Supporting health among young men who have sex with men and transgender women with HIV: Lessons learned from implementing the weCare intervention. *Health Promot Pract.* 2020;21(5):755-763.
- 13. Tanner AE, Dowshen N, Philbin MM, et al. An intervention for the transition from pediatric or adolescent to adult-oriented HIV care: Protocol for the development and pilot implementation of iTransition. *JMIR Res Protoc.* 2021;10(4):e24565.
- 14. Medich M, Swendeman DT, Comulada WS, Kao UH, Myers JJ, Brooks RA, Special Projects of National Significane Social Media Initiative Study Group. Promising approaches for engaging youth and young adults living with HIV in HIV primary care using social media and mobile technology interventions: Protocol for the SPNS Social Media Initiative. *JMIR Res Protoc.* 2019;8(1):e10681.
- 15. Rhodes SD, Hergenrather KC, Bloom FR, Leichliter JS, Montano J. Outcomes from a community-based, participatory lay health adviser HIV/STD prevention intervention for recently arrived immigrant Latino men in rural North Carolina. *AIDS Educ Prev.* 2009;21(5 Suppl):103-108.
- 16. Rhodes SD, Leichliter JS, Sun CJ, Bloom FR. The HoMBReS and HoMBReS Por un Cambio interventions to reduce HIV disparities among immigrant Hispanic/Latino men. *MMWR Morb Mortal Wkly Rep.* 2016;65(1):51-56.
- 17. Martinez O, Roth AM, Kelle G, Downs M, Rhodes SD. Adaptation and implementation of HoMBReS: A community-level, evidence-based HIV behavioral intervention for heterosexual Latino men in the midwestern United States. *AIDS Educ Prev.* 2014;26(1):68-80.
- 18. Rhodes SD, Alonzo J, Mann L, et al. Enhancement of a locally developed HIV prevention intervention for Hispanic/Latino MSM: A partnership of community-based organizations, a university, and the Centers for Disease Control and Prevention *AIDS Educ Prev.* 2015;27(4):312-332.

- 19. Rhodes SD, Daniel J, Alonzo J, Duck S, Garcia M, Downs M, Hergenrather KC, Alegria-Ortega J, Miller C, Boeving Allen A, Gilbert PA, Marsiglia FF. A systematic community-based participatory approach to refining an evidence-based community-level intervention: The HOLA intervention for Latino men who have sex with men. *Health Promot Pract.* 2013;14(4):607-616.
- 20. Sun CJ, Garcia M, Mann L, Alonzo J, Eng E, Rhodes SD. Latino sexual and gender identity minorities promoting sexual health within their social networks: process evaluation findings from a lay health advisor intervention. *Health Promot Pract.* 2015;16(3):329-337.
- 21. Rhodes SD, Kelley C, Simán F, Cashman R, Alonzo J, McGuire J, Wellendorf T, Hindshaw K, Boeving Allen A, Downs M, Brown M, Martinez O, Duck S, Reboussin B. Using community-based participatory research (CBPR) to develop a community-level HIV prevention intervention for Latinas: A local response to a global challenge. *Womens Health Issues*. 2012;22(3):293-301.
- 22. Painter TM, Organista KC, Rhodes SD, Sañudo FM. Interventions to prevent HIV and other sexually transmitted diseases among Latino migrants. In: Organista KC, ed. *HIV Prevention with Latinos: Theory, Research, and Practice*. New York, NY: Oxford; 2012:351-381.
- 23. Sun CJ, Mann L, Eng E, Downs M, Rhodes SD. Once a Navegante, always a Navegante: Latino men sustain their roles as lay health advisors to promote general and sexual health to their social network. *AIDS Education and Prevention.* 2015;27(5):465-473.
- 24. Rhodes SD, Alonzo J, Mann-Jackson L, Song EY, Tanner AE, Garcia M, Smart BD, Baker LS, Eng E, Reboussin BA. A peer navigation intervention to prevent HIV among mixed immigrant status Latinx GBMSM and transgender women in the United States: Outcomes, perspectives and implications for PrEP uptake *Health Educ Res.* 2020;35(3):165-178.
- 25. Aronson RE, Rulison KL, Graham LF, McCoy Pulliam R, McGee WL, Labban JD, Dingman D, Rhodes SD. Brothers Leading Healthy Lives: Outcomes from the pilot testing of a culturally and contextually congruent HIV prevention intervention for black male college students. *AIDS Educ Prev.* 2013;25(5):376-393.
- 26. Rhodes SD, Mann L, Alonzo J, Downs M, Abraham C, Miller C, Stowers J, Ramsey B, Simán FM, Song E, Vissman AT, Eng E, Reboussin BA CBPR to prevent HIV within ethnic, sexual, and gender minority communities: Successes with long-term sustainability. In: Rhodes SD, ed. *Innovations in HIV Prevention Research and Practice through Community Engagement*. New York, NY: Springer; 2014:135-160.
- 27. Rhodes SD, Mann-Jackson L, Alonzo J, Nall J, Siman FM, Song EY, Garcia M, Tanner AE, Eng E. Harnessing "Scale-Up and Spread" to support community uptake of the HoMBReS por un Cambio intervention for Spanish-Speaking men: Implementation science lessons learned by a CBPR partnership. *Am J Mens Health*. 2020;14(4):1557988320938939.
- 28. Eng E, Rhodes SD, Parker EA. Natural helper models to enhance a community's health and competence. In: DiClemente RJ, Crosby RA, Kegler MC, eds. *Emerging Theories in Health Promotion Practice and Research*. Vol 2. San Francisco, CA: Jossey-Bass; 2009:303-330.
- 29. Rhodes SD, McCoy TP, Tanner AE, et al. Using social media to increase HIV testing among gay and bisexual men, other MSM, and transgender persons: Outcomes from a randomized community trial. *Clin Infect Dis.* 2016;62(11):1450-1453.
- 30. Rhodes SD, Vissman AT, Stowers J, Miller C, McCoy TP, Hergenrather KC, Wilkin AM, Reece M, Bachmann LH, Ore A, Ross MW, Hendrix E, Eng E. A CBPR partnership increases HIV testing among men who have sex with men (MSM): Outcome findings from a pilot test of the CyBER/testing Internet intervention. *Health Educ Behav.* 2011;38(3):311-320.
- 31. Sun CJ, Stowers J, Miller C, Bachmann LH, Rhodes SD. Acceptability and feasibility of using established geosocial and sexual networking mobile applications to promote HIV and STD testing among men who have sex with men. *AIDS and Behavior*. 2015;19(3):543-552.
- 32. Jenkins Hall W, Sun CJ, Tanner AE, Mann L, Stowers J, Rhodes SD. HIV-prevention opportunities with GPS-based social and sexual networking applications for men who have sex with men. *AIDS Educ Prev.* 2017;29(1):38-48.

- 33. Van Dyke ME, Mendoza MCB, Li W, et al. Racial and ethnic disparities in COVID-19 incidence by age, sex, and period among persons aged <25 years 16 U.S. jurisdictions, January 1-December 31, 2020. *MMWR Morb Mortal Wkly Rep.* 2021;70(11):382-388.
- 34. Martinez AD, Rhodes SD. Introduction: Disentangling language and the social determinants of Latinx health in the United States. In: Martinez AD, Rhodes SD, eds. *New and Emerging Issues in Latinx Health*. Switzerland: Springer; 2020:1-15.
- 35. Ornelas IJ, Yamanis TJ, Ruiz RA. The health of undocumented Latinx immigrants: What we know and future directions. *Annu Rev Public Health*. 2020;41:289-308.
- 36. Demographic Trends of COVID-19 Cases and Deaths in the US Reported to CDC. 2021. https://covid.cdc.gov/covid-data-tracker/#demographics.
- 37. Guynn J, Marcos CM. COVID-19 crisis: Vaccine Conspiracy Theories, Hoaxes in Spanish Targeting Hispanic Community Breed Fear, Hesitancy. *USA Today*. 2021.
- 38. Ajazeera A. COVID Vaccine Scarcity and Fake Doses Hamper Efforts in Americas. 2021. https://www.aljazeera.com/news/2021/4/21/covid-vaccine-scarcity-and-fake-doses-hamper-efforts-in-americas
- 39. BBC News. Coronavirus: Pfizer Confirms Fake Versions of Vaccine in Poland and Mexico. 2021. https://www.bbc.com/news/world-56844149
- 40. Hispanic League. *Reflection & Metrics for Greater Impact*. Winston-Salem, NC: Hispanic League. 2021.
- 41. Laurencin CT, Wu ZH, McClinton A, Grady JJ, Walker JM. Excess deaths among Blacks and Latinx compared to Whites during Covid-19. *J Racial Ethn Health Disparities*. 2021;8(3):783-789.
- 42. Moyce S, Velazquez M, Claudio D, et al. Exploring a rural Latino community's perception of the COVID-19 pandemic. *Ethn Health.* 2021;26(1):126-138.
- 43. Pan D, Sze S, Minhas JS, et al. The impact of ethnicity on clinical outcomes in COVID-19: A systematic review. *EClinicalMedicine*. 2020;23:100404.
- 44. Wilder JM. The disproportionate impact of COVID-19 on racial and ethnic minorities in the United States. *Clin Infect Dis.* 2020;72(4):707-709.
- 45. Marsiglia FF, Kulis S. Diversity, Oppression, and Change. Chicago, IL: Lyceum; 2009.
- 46. Camacho-Rivera M, Gonzalez CJ, Morency JA, Blake KD, Calixte R. Heterogeneity in trust of cancer information among Hispanic Adults in the United States: An analysis of the Health Information National Trends Survey. *Cancer Epidemiol Biomarkers Prev.* 2020;29(7):1348-1356.
- 47. Singer MA, Velez MG, Rhodes SD, Linton JM. Discrimination against mixed-status families and its health impact on Latino children. *J Appl Res Child*. 2018;10(1):6.
- 48. Budiman A, Tamir C, Mora L, Noe-Bustamante L. *Facts on U.S. Immigrants, 2018.* Washington, DC: Pew Research Center. 2020.
- 49. Vines AI, Hunter JC, Carlisle VA, Richmond AN. Prostate Cancer Ambassadors: Process and outcomes of a prostate cancer informed decision-making training program. *Am J Mens Health*. 2016;11(1):54-62.
- 50. Rhodes SD, Daniel J, Alonzo J, et al. A snapshot of how Latino heterosexual men promote sexual health within their social networks: Process evaluation findings from an efficacious community-level intervention. *AIDS Educ Prev.* 2012;24(6):514-526.
- 51. Flora PK, Bender JL, Miller AS, et al. A core competency framework for prostate cancer peer navigation. *Support Care Cancer*. 2019;28(6):2605-2614.
- 52. Herce ME, Muyoyeta M, Topp SM, Henostroza G, Reid SE. Coordinating the prevention, treatment, and care continuum for HIV-associated tuberculosis in prisons: A health systems strengthening approach. *Curr Opin HIV AIDS*. 2018;13(6):492-500.
- 53. Cunningham WE, Weiss RE, Nakazono T, et al. Effectiveness of a peer navigation intervention to sustain viral suppression among HIV-positive men and transgender women released from jail: The LINK LA Randomized Clinical Trial. *JAMA Intern Med.* 2018;178(4):542-553.

- 54. Cabral HJ, Davis-Plourde K, Sarango M, Fox J, Palmisano J, Rajabiun S. Peer Support and the HIV continuum of care: Results from a multi-site randomized clinical trial in three urban clinics in the United States. *AIDS Behav.* 2018;22(8):2627-2639.
- 55. Corrigan PW, Pickett S, Schmidt A, et al. Peer navigators to promote engagement of homeless African Americans with serious mental illness in primary care. *Psychiatry Res.* 2017;255:101-103.
- 56. Adams JA, Whiteman K, McGraw S. Reducing missed appointments for patients with HIV: An evidence-based approach. *J Nurs Care Qual.* 2020;35(2):165-170.
- 57. Goodman-Meza D, Shoptaw S, Weiss RE, et al. Methamphetamine use drives decreases in viral suppression for people living with HIV released from a large municipal jail: Results of the LINK LA clinical trial. *Drug Alcohol Depend.* 2019;202:178-184.
- 58. Oliver CD, Rebeiro PF, Shepherd BE, et al. Clinic-level factors associated with retention in care among people living with HIV in a multi-site United States cohort, 2010-2016. *Clin Infect Dis.* 2019.
- 59. Samuels EA, Bernstein SL, Marshall BDL, Krieger M, Baird J, Mello MJ. Peer navigation and takehome naloxone for opioid overdose emergency department patients: Preliminary patient outcomes. *J Subst Abuse Treat.* 2018:94:29-34.
- 60. Wilson EC, Turner C, Arayasirikul S, et al. HIV care engagement among trans women of color in San Francisco Bay area demonstration projects: Findings from the Brandy Martell Project and TransAccess. *AIDS Behav.* 2019.
- 61. Rebchook G, Keatley J, Contreras R, et al. The Transgender Women of Color Initiative: Implementing and evaluating innovative interventions to enhance engagement and retention in HIV care. *Am J Public Health.* 2017;107(2):224-229.
- 62. Rhodes SD, Alonzo J, Mann L, et al. Novel approaches to HIV prevention and sexual health promotion among Guatemalan gay and bisexual men, MSM, and transgender persons *AIDS Education and Prevention*. 2014;26(4):345-361.
- 63. Rhodes SD, Foley KL, Zometa CS, Bloom FR. Lay health advisor interventions among Hispanics/Latinos: A qualitative systematic review. *Am J Prev Med.* 2007;33(5):418-427.
- 64. Vissman AT, Eng E, Aronson RE, et al. What do men who serve as lay health advisors really do?: Immigrant Latino men share their experiences as *Navegantes* to prevent HIV. *AIDS Education and Prevention*. 2009;21(3):220-232.
- 65. Hudnut-Beumler J, Po'e E, Barkin S. The use of social media for health promotion in Hispanic populations: A scoping systematic review. *JMIR Public Health Surveill*. 2016;2(2):e32.
- 66. Chou WS, Gaysynsky A, Trivedi N, Vanderpool RC. Using social media for health: National data from HINTS 2019. *J Health Commun*. 2021;26(3):184-193.
- 67. Rodriquez EJ, Pérez-Stable EJ. The time is now for eHealth research with Latinos. *Am J Public Health*. 2017;107(11):1705-1707.
- 68. Mueller NT, Noone AM, Luta G, Wallington SF, Huerta EE, Mandelblatt JS. Information channels associated with awareness of human papillomavirus infections and vaccination among Latino immigrants from safety net clinics. *J Immigr Minor Health*. 2012;14(1):183-188.
- 69. Victorson D, Banas J, Smith J, et al. eSalud: Designing and implementing culturally competent ehealth research with latino patient populations. *Am J Public Health*. 2014;104(12):2259-2265.
- 70. Mann-Jackson L, Alonzo J, Garcia M, Trent S, Bell J, Horridge DN, Rhodes SD. Using community-based participatory research to address STI/HIV disparities and social determinants of health among young GBMSM and transgender women of colour in North Carolina, USA. *Health Soc Care Community*. Epub ahead of print.
- 71. Anderson M, Kumar M. *Digital Divide Persists Even as Lower-Income Americans Make Gains in Tech Adoption*. Washington, DC: Pew Research Center. 2019.
- 72. Muessig KE, Nekkanti M, Bauermeister J, Bull S, Hightow-Weidman LB. A systematic review of recent smartphone, Internet and Web 2.0 interventions to address the HIV continuum of care. *Curr HIV/AIDS Rep.* 2015;12(1):173-190.
- 73. Cervantes L, Martin M, Frank MG, et al. Experiences of Latinx individuals hospitalized for COVID-19: A qualitative study. *JAMA Netw Open.* 2021;4(3):e210684.

- 74. Campos-Castillo C, Anthony D. Racial and ethnic differences in self-reported telehealth use during the COVID-19 pandemic: a secondary analysis of a US survey of internet users from late March. *J Am Med Inform Assoc.* 2021;28(1):119-125.
- 75. Perrin A, Anderson MB. Share of U.S. Adults Using Social Media, Including Facebook, Is Mostly Unchanged Since 2018. 2019.
- 76. Perrin A, Turner E. Smartphones Help Blacks, Hispanics Bridge Some But Not All Digital Gaps with Whites. Washington, DC: Pew Research Center. 2019.
- 77. Pew Research Center. Mobile fact sheet. Washington, DC: Pew Research Center;2019.
- 78. Duggan M, Ellison NB, Lampe C, Lenhart A, Madden M. *Social Media Update*. Washington, DC: Pew Research Center. 2015. Available at: http://www.pewinternet.org/2015/01/09/social-media-update-2014/.
- 79. Northcott C, Curtis R, Bogomolova S, et al. Evaluating the effectiveness of a physical activity social media advertising campaign using Facebook, Facebook Messenger, and Instagram. *Transl Behav Med*. 2021;11(3):870-881.
- 80. Young SD, Holloway I, Jaganath D, Rice E, Westmoreland D, Coates T. Project HOPE: online social network changes in an HIV prevention randomized controlled trial for African American and Latino men who have sex with men. *Am J Public Health*. 2014;104(9):1707-1712.
- 81. Williams CB, LaCoursiere DY, Talavera GA, Gahagan S. A feasibility study to promote optimal weight in first time pregnant mothers and their babies: Lessons learned in a US-Mexico border community. *Matern Child Health J.* 2019;23(5):578-584.
- 82. Bull S, Walker T, Levine D. Communities and technology: Enhancements in HIV-prevention research and practice among adolescents and young adults. In: Rhodes SD, ed. *Innovations in HIV Prevention Research and Practice through Community Engagement*. New York, NY: Springer; 2014:183-214.
- 83. Bull SS. Sexually transmitted disease prevention campaigns in the 21st century: new frontiers in social media. *Sex Transm Dis.* 2014;41(3):158-160.
- 84. Cole-Lewis H, Kershaw T. Text messaging as a tool for behavior change in disease prevention and management. *Epidemiol Rev.* 2010;32(1):56-69.
- 85. Mbuagbaw L, Mursleen S, Lytvyn L, Smieja M, Dolovich L, Thabane L. Mobile phone text messaging interventions for HIV and other chronic diseases: An overview of systematic reviews and framework for evidence transfer. *BMC Health Serv Res.* 2015;15(1):33.
- 86. Christopoulos KA, Riley ED, Tulsky J, et al. A text messaging intervention to improve retention in care and virologic suppression in a U.S. urban safety-net HIV clinic: study protocol for the Connect4Care (C4C) randomized controlled trial. *BMC Infect Dis.* 2014;14(1):3849.
- 87. Horvath T, Azman H, Kennedy GE, Rutherford GW. Mobile phone text messaging for promoting adherence to antiretroviral therapy in patients with HIV infection. *Cochrane Database Syst Rev.* 2012;3:CD009756.
- 88. Ramirez M, Wu S, Beale E. Designing a text messaging intervention to improve physical activity behavior among low-income Latino patients with diabetes: A discrete-choice experiment, Los Angeles, 2014-2015. *Prev Chronic Dis.* 2016;13:E171.
- 89. Silverman-Lloyd LG, Dominguez Cortez J, Godage SK, et al. Immigrant Latino parents demonstrated high interactivity with pediatric primary care text messaging intervention. *Mhealth.* 2020;6:45.
- 90. Fareed N, Swoboda CM, Jonnalagadda P, Walker DM, Huerta TR. Differences between races in health information seeking and trust over time: Evidence from a cross-sectional, pooled analyses of HINTS data. *Am J Health Promot.* 2021;35(1):84-92.
- 91. Kelly BJ, Southwell BG, McCormack LA, et al. Predictors of willingness to get a COVID-19 vaccine in the U.S. *BMC Infect Dis.* 2021;21(1):338.
- 92. Kearney A, Lopes L, Brodie M. *Vaccine Hesitancy Among Hispanic Adults*. San Francisco, CA: Kaiser Family Foundation. 2021.
- 93. Rhodes SD. Demonstrated effectiveness and potential of CBPR for preventing HIV in Latino populations. In: Organista KC, ed. *HIV Prevention with Latinos: Theory, Research, and Practice*. New York, NY: Oxford; 2012:83-102.

- 94. Rhodes SD. Authentic engagement and community-based participatory research for public health and medicine. In: Rhodes SD, ed. *Innovations in HIV Prevention Research and Practice through Community Engagement*. New York, NY: Springer; 2014:1-10.
- 95. Rhodes SD, Alonzo J, Mann L, Siman FM, Garcia M, Abraham C, Sun CJ. Using photovoice, Latina transgender women identify priorities in a new immigrant-destination state. *Int J Transgend*. 2015;16(2):80-96.
- 96. Rhodes SD, Duck S, Alonzo J, Daniel J, Aronson RE. Using community-based participatory research to prevent HIV disparities: Assumptions and opportunities identified by The Latino Partnership. *J Acquir Immune Defic Syndr*. 2013;63(Supplement 1):S32-S35.
- 97. Rhodes SD, Eng E, Hergenrather KC, et al. Exploring Latino men's HIV risk using community-based participatory research. *Am J Health Behav.* 2007;31(2):146-158.
- 98. Rhodes SD, Hergenrather KC, Aronson RE, Bloom F, Felizzola J, Wolfson M, Vissman AT, Alonzo J, Boeving Allen A, Montano J, McGuire J. Latino men who have sex with men and HIV in the rural south-eastern USA: Findings from ethnographic in-depth interviews. *Cult Health Sex.* 2010;12(7):797-812.
- 99. Rhodes SD, Hergenrather KC, Duncan J, Ramsey B, Yee LJ, Wilkin AM. Using community-based participatory research to develop a chat room-based HIV prevention intervention for gay men. *Prog Community Health Partnersh.* 2007;1(2):175-184.
- 100. Rhodes SD, Hergenrather KC, Vissman AT, Stowers J, Davis AB, Hannah A, Alonzo J, Marsiglia FF. Boys must be men, and men must have sex with women: A qualitative CBPR study to explore sexual risk among African American, Latino, and white gay men and MSM. *Am J Mens Health*. 2011;5(2):140-151.
- 101. Rhodes SD, Mann L, Siman FM, Alonzo J, Vissman AT, Nall J, Tanner AE. ENGAGED for CHANGE: An innovative community-based participatory research strategy to intervention development. In: Wallerstein N, Duran B, Oetzel J, Minkler M, eds. *Community-Based Participatory Research for Health*. 3 ed. San Francisco, CA: Jossey-Bass; 2017.
- 102. Rhodes SD, McCoy TP, Vissman AT, DiClemente RJ, Duck S, Hergenrather KC, Foley KL, Alonzo J, Bloom F, Eng E. A randomized controlled trial of a culturally congruent intervention to increase condom use and HIV testing among heterosexually active immigrant Latino men. *AIDS Behav*. 2011;15(8):1764-1775.
- 103. Rhodes SD, Tanner AE, Mann-Jackson L, Alonzo J, et al. Promoting community and population health in public health and medicine: A stepwise guide to initiating and conducting community-engaged research. *J Health Dispar Res Pract.* 2018;11(3):16-31.
- 104. Rhodes SD, Tanner AE, Mann-Jackson L, Alonzo J, et al. Community-engaged research as an approach to expedite advances in HIV prevention, care, and treatment: A call to action. *AIDS Educ Prev.* 2018;30(3):243-253.
- 105. Mann L, Simán FM, Downs M, Sun CJ, Urquieta de Hernandez B, Garcia M, Alonzo J, Lawlor E, Rhodes SD. Reducing the impact of immigration enforcement policies to ensure the health of North Carolinians: Statewide community-level recommendations. *NC Med J.* 2016;77(4):240-246.
- 106. A National Institute of Nursing Research Workshop. *State of Rural Health Disparities: Research Gaps and Recommendations*. Bethesda, MD: Available at: https://www.ninr.nih.gov/sites/files/docs/2018-State-of-Rural-Health-Disparities-NINR-Workshop-508c.pdf. 2018.
- 107. Agency for Healthcare Research and Quality. *Community-Based Participatory Research*. Rockville, MD: Available at: http://www.ahrq.gov/about/cbpr/cbpr. 2002.
- 108. Bogart LM, Uyeda K. Community-based participatory research: Partnering with communities for effective and sustainable behavioral health interventions. *Health Psychol.* 2009;28(4):391-393.
- 109. Burhansstipanov L, Christopher S, Schumacher SA. Lessons learned from community-based participatory research in Indian country. *Cancer Control*. 2005;12 Suppl 2:70-76.
- 110. Cacari-Stone L, Wallerstein N, Garcia AP, Minkler M. The promise of community-based participatory research for health equity: A conceptual model for bridging evidence with policy. *Am J Public Health*. 2014;104(9):1615-1623.

- 111. Cashman SB, Adeky S, Allen AJ,... Rhodes SD, et al. The power and the promise: Working with communities to analyze data, interpret findings, and get to outcomes. *Am J Public Health*. 2008;98(8):1407-1417.
- 112. Clements-Nolle K, Bachrach AM. CBPR within a hidden population: The Transgender Community Health Project a decade later. In: Minkler M, Wallerstein N, eds. *Community-based Participatory Research for Health*. 2 ed. San Francisco, CA: Wiley; 2008:137-151.
- 113. Leshner AI, Terry SF, Schultz AM, Liverman CT, eds. *The CTSA Program at NIH: Opportunities for Advancing Clinical and Translational Research*. Institute of Medicine of the National Academies. 2013.
- 114. Institute of Medicine. *Unequal Treatment: Confronting Racial and Ethnic Disparities in Health Care.* Washington, DC: National Academy Press. 2003.
- 115. Rhodes SD, Daniel-Ulloa J, Wright SS, Mann-Jackson L, et al. Critical elements of community engagement to address disparities and related social determinants of health: The Centers of Disease Control and Prevention Community Approaches to Reducing Sexually Transmitted Disease initiative. *Sex Transm Dis.* 2021;48(1):49-55.
- 116. Irby MB, Moore KR, Hamlin D, Brown O, trejo D, Summers P, Daniel S, Skelton JA, Lischke M, Rhodes SD. Building bridges between a community and an academic medical center via community tours. *J Clin Transl Sci.* 2020;4(4):294-300.
- 117. Irby MB, Moore KR, Mann-Jackson L,... Rhodes SD. Community-engaged research: Common themes and needs identified by investigators and research teams at an emerging academic learning health system. *Int J Environ Res Public Health*. 2021;18(8).
- 118. Dilley JR, Moore JB, Summers P,... Bertoni AG. A citizen science approach to determine physical activity patterns and demographics of greenway users in Winston-Salem, North Carolina. *Int J Environ Res Public Health*. 2019;16(17).
- 119. Minkler M. Linking science and policy through community-based participatory research to study and address health disparities. *Am J Public Health*. 2010;100 Suppl 1:S81-87.
- 120. Wallerstein N, Duran B. Community-based participatory research contributions to intervention research: The intersection of science and practice to improve health equity. *Am J Public Health*. 2010;100 Suppl 1:S40-46.
- 121. Caldwell WB, Reyes AG, Rowe Z, Weinert J, Israel BA. Community partner perspectives on benefits, challenges, facilitating factors, and lessons learned from community-based participatory research partnerships in Detroit. *Prog Community Health Partnersh.* 2015;9(2):299-311.
- 122. Wolfson M, Wagoner KG, Rhodes SD, et al. Coproduction of research questions and research evidence in public health: The study to prevent teen drinking parties. *Biomed Res Int.* 2017;3639596.
- 123. Samuel CA, Lightfoot AF, Schaal J, et al. Establishing new community-based participatory research partnerships using the community-based participatory research Charrette Model: Lessons from the Cancer Health Accountability for Managing Pain and Symptoms Study. *Prog Community Health Partnersh*. 2018;12(1):89-99.
- 124. Rhodes SD, Alonzo J, Mann L, Song EY, Tanner AE, Arellano JE, Rodriguez-Celedon R, Garcia M, Freeman A, Reboussin BA, Painter TM. Small-group randomized controlled trial to increase condom use and HIV testing among Hispanic/Latino gay, bisexual, and other men who have sex with men. *Am J Public Health*. 2017;107(6):969-976.
- 125. Rhodes SD. Community-based participatory research. In: Blessing JD, Forister. JG, eds. *Introduction to Research and Medical Literature for Health Professionals.* 3 ed. Burlington, MA: Jones & Bartlett; 2013:167-187.
- 126. Rhodes SD, Alonzo J, Mann Jackson L, Tanner AE, Vissman AT, Martinez O, Rodrigo-Celedon R, Garcia JM, Arellano JE, Song EY, Eng E, Rebossin BA. Selling the product: Strategies to increase recruitment and retention of Spanish-speaking Latinos in biomedical research. *J Clin Transl Sci.* 2018;2(3):147-155.

- 127. Israel BA, Krieger J, Vlahov D, et al. Challenges and facilitating factors in sustaining community-based participatory research partnerships: lessons learned from the Detroit, New York City and Seattle Urban Research Centers. *J Urban Health*. 2006;83(6):1022-1040.
- 128. Israel BA, Lichtenstein R, Lantz P, et al. The Detroit Community-Academic Urban Research Center: Development, implementation, and evaluation. *J Public Health Manag Pract.* 2001;7(5):1-19.
- 129. Israel BA, Schulz AJ, Parker EA, Becker AB. Review of community-based research: Assessing partnership approaches to improve public health. *Annu Rev Public Health*. 1998;19:173-202.
- 130. Mann-Jackson L, Song EY, Tanner AE, Alonzo J, Linton JM, Rhodes SD. The health impact of experiences of discrimination, violence, and immigration enforcement among Latino men in a new settlement state. *Am J Mens Health*. 2018:1557988318785091.
- 131. Tanner AE, Chambers BD, Philbin MM, et al. The intersection between women's reproductive desires and HIV care providers' reproductive health practices: A mixed methods analysis. *Matern Child Health J.* 2018;22(9):1233-1239.
- 132. Rhodes SD, Mann L, Simán FM, Song E, Alonzo J, Lawlor E, Martinez O, Sun CJ, O'Brien MC, Rebossin BA, Hall MA. The impact of local immigration enforcement policies on the health of immigrant Hispanics/Latinos in the United States. *Am J Public Health*. 2015;105(2):329-337.
- 133. Rhodes SD, Mann-Jackson L, Song EY, Wolfson M, Filindra A, Hall MA. Laws and policies related to the health of US immigrants: A policy scan. *Health Behav Policy Rev.* 2020;7(4):314-324.
- 134. Rhodes SD, Kuhns LM, Alexander J, Alonzo J, Bessler P, Courtenay-Quirk C, Denson DJ, Evans K, Galindo CA, Garofalo R, Gelaude D, Hotton AL, Johnson AK, Mann-Jackson L, Muldoon A, Ortiz R, Paul JL, Perlaoff J, Pleasant K, Reboussin BA, Refugio Aviles L, Song EY, Tanner AE, Trent S. Evaluating homegrown interventions to promote PrEP among racially/ethnically diverse transgender women in the United States: A unique CDC initiative. *AIDS Educ Prev.* 2021;33(4): In press.
- 135. Rhodes SD, Hergenrather KC, Duncan J, et al. A pilot intervention utilizing Internet chat rooms to prevent HIV risk behaviors among men who have sex with men. *Public Health Reports*. 2010;125(Supplement 1):29-37.
- 136. Rhodes SD, Hergenrather KC, Yee LJ, Ramsey B. Comparing MSM in the southeastern United States who participated in an HIV prevention chat room-based outreach intervention and those who did not: how different are the baseline HIV-risk profiles? *Health Educ Res.* 2008;23(1):180-190.
- 137. Rhodes SD, Hergenrather KC, Montano J, et al. Using community-based participatory research to develop an intervention to reduce HIV and STD infections among Latino men. *AIDS Educ Prev.* 2006;18(5):375-389.
- 138. Tanner AE, Reboussin BA, Mann L, Ma A, Song E, Alonzo J, Rhodes SD. Factors influencing healthcare access perceptions and care-seeking behaviors of Latino sexual minority men and transgender individuals: HOLA intervention baseline findings. *J Health Care Poor Underserved*. 2014;25(4):1679-1697.
- 139. US Census Bureau. http://www.census.gov/2021.
- 140. Seña AC, Weber DJ. From health disparities to hotspots to public health strategies: The impact of the COVID-19 pandemic in North Carolina. *N C Med J.* 2021;82(1):37-42.
- 141. DuBard CA, Gizlice Z. Language spoken and differences in health status, access to care, and receipt of preventive services among US Hispanics. *Am J Public Health*. 2008;98(11):2021-2028.
- 142. Ndugga N, Pham O, Hill L, Artiga S, Parker N. *Latest Data on COVID-19 Vaccinations Race/Ethnicity*. 2021.
- 143. Rhodes SD, Malow RM, Jolly C. Community-based participatory research: a new and not-so-new approach to HIV/AIDS prevention, care, and treatment. *AIDS Educ Prev.* 2010;22(3):173-183.
- 144. Charmaz K. Constructing Grounded Theory: A Practical Guide through Qualitative Analysis. London: Sage. 2006.
- 145. Coffey A, Atkinson P. Making Sense of Qualitative Data. Thousand Oaks, CA: Sage; 1996.
- 146. Creswell JW. *Qualitative Inquiry and Research Design: Choosing Among Five Traditions*. Thousand Oaks, CA: Sage. 1998.

- 147. Fontana A, Frey JH. Interviewing: The art of science. In: Denzin NK, Lincoln YS, eds. *Collecting and Interpreting Qualitative Materials*. Thousand Oaks, CA: Sage. 1998:47-78.
- 148. Lincoln YS, Guba EG. Paradigmatic controversies, contradictions, and emerging confluences. In: Denzin NK, Lincoln YS, eds. *The Handbook of Qualitative Research*. 2 ed. Thousand Oaks: Sage. 2000:163-188.
- 149. Morse J. Designing funded qualitative research. In: Denzen N, Lincoln Y, eds. *Handbook of Qualitative Research*. Thousand Oaks, CA: Sage. 1994:220-235.
- 150. Patton MQ. *Qualitative Evaluation and Research Methods*. Second edition ed. Newbury Park, CA: Sage. 1990.
- 151. Rhodes SD, Sy FS. Effectively confronting the COVID-19 pandemic: Critical lessons from HIV prevention, care, and treatment and innovative strategies to conduct community-based and community-engaged research safely. *AIDS Educ Prev.* 2020;32(6):455-471.
- 152. Resnicow K, Baranowski T, Ahluwalia JS, Braithwaite RL. Cultural sensitivity in public health: Defined and demystified. *Ethn Dis.* 1999;9(1):10-21.
- 153. Munn P, Drever E. *Using Questionnaires in Small-scale Research: A Teacher's Guide*. Glasgow, Scotland: Scottish Council For Research In Education; 1995.
- 154. Rubin HJ, Rubin IS. *Qualitative Data: The art of hearing data*. 2 ed. Thousand Oaks, CA: Sage; 2005
- 155. Spradley JP. The Ethnographic Interview. New York, NY: Holt, Rinehart, & Winston. 1979.
- 156. Merriam S. *Qualitative Research and Case Study Applications in Education*. San Francisco, CA: Jossey-Bass. 1998.
- 157. Glaser BG, Strauss AL. *The Discovery of Grounded Theory: Strategies for Qualitative Research.* Chicago, IL: Aldine. 1967.
- 158. McCabe JM, Tanner AE, Heiman J. The impact of gender expectations on meanings of sex and sexuality: Results from a cognitive interview study. *Sex Roles*. 2010;63(2):252-263.
- 159. Goetz JP, LeCompte MD. *Ethnography and Qualitative Design in Educational Research*. Orlando, FL: Academic Press Inc. 1984.
- 160. Miles AM, Huberman MM. *Qualitative Data Analysis: An Expanded Sourcebook.* 2nd ed. Thousand Oaks, CA: Sage. 1994.
- 161. Rhodes SD, Alonzo J, Mann L, et al. The ecology of sexual health of sexual minorities in Guatemala City. *Health Promot Int.* 2015;30(4):832-842.
- 162. Shibusawa T, Lukens E. Analyzing qualitative data in a cross-language context: A collaborative model. In: Padgett DK, ed. *The Qualitative Research Experience*. Belmont, CA: Wadsworth/Thomson Learning. 2004:175-186.
- 163. Silverman D. *Interpreting qualitative data: Methods for Analysing Talk, Text and Interaction.* London: Sage. 2001.
- 164. Strauss A, Corbin J. *Basics of Qualitative Research*. 2 ed. Thousand Oaks, CA: Sage Publications. 1998.
- 165. Streng JM, Rhodes SD, Ayala GX, Eng E, Arceo R, Phipps S. Realidad Latina: Latino adolescents, their school, and a university use photovoice to examine and address the influence of immigration. *J Interprof Care*. 2004;18(4):403-415.
- 166. Eng E, Moore KS, Rhodes SD, et al. Insiders and outsiders assess who is "the community": Participant observation, key informant interview, focus group interview, and community forum. In: Israel BA, Eng E, Schulz AJ, Parker E, eds. *Methods for Conducting Community-Based Participatory Research for Health*. San Francisco, CA: Jossey-Bass; 2005:77-100.
- 167. Rhodes SD, Duck S, Alonzo J, Downs M, Aronson RE. Intervention trials in community-based participatory research. In: Blumenthal D, DiClemente RJ, Braithwaite RL, Smith S, eds. *Community-Based Participatory Research: Issues, Methods, and Translation to Practice.* New York: Springer 2013:157-180.
- 168. Bandura A. *Social Foundations of Thought and Action: A Social Cognitive Theory*. Englewood Cliffs: Prentice-Hall; 1986.

- 169. Freire P. Education for Critical Consciousness. New York, NY: Seabury Press; 1973.
- 170. Wills TA. Supportive functions of interpersonal relationships. In: Cohen S, Syme L, eds. *Social Support and Health*. Orlando, FL: Academic Press. 1985:61-82.
- 171. Chou W-YS, Burgdorf CE, Gaysynsky A, Hunter CM. *COVID-19 Vaccination Communication: Applying Behavioral and Social Science to Address Vaccine Hesitancy and Foster Vaccine Confidence.* Bethesda, MD: National Institutes of Health. 2020.
- 172. RADx-UP. Resource Library. https://www.kumc.edu/school-of-medicine/population-health/radxup/resource-library.html. Published 2021. Accessed May 30, 2021.
- 173. Rhodes SD, Mann-Jackson L, Alonzo J, Siman FM, Vissman AT, Nall J, Abraham C, Aronson RE, Tanner AE. The ENGAGED for CHANGE process for developing interventions to reduce health disparities. *AIDS Educ Prev.* 2017;29(6):491-502.
- 174. Young S. Healthy behavior change in practical settings. *Perm J.* 2014;18(4):89-92.
- 175. Rowland SP, Fitzgerald JE, Holme T, Powell J, McGregor A. What is the clinical value of mHealth for patients? *NPJ Digit Med.* 2020;3:4.
- 176. Pozzana I, Ferrara E. Measuring Bot and Human Behavioral Dynamics. Available at: https://arxivorg/pdf/180204286pdf. 2018.
- 177. Navarro AM, Senn KL, McNicholas LJ, Kaplan RM, Roppe B, Campo MC. Por La Vida model intervention enhances use of cancer screening tests among Latinas. *Am J Prev Med.* 1998;15(1):32-41.
- 178. Dunn TJ, Baguley T, Brunsden V. From alpha to omega: A practical solution to the pervasive problem of internal consistency estimation. *Br J Psychol.* 2014;105(3):399-412.
- 179. Friedman LM, Furberg CD, DeMets DL. *Fundamentals of Clinical Trials*. 3 ed. New York, NY: Springer-Verlag; 1998.
- 180. Leyrat C, Caille A, Foucher Y, Giraudeau B. Propensity score to detect baseline imbalance in cluster randomized trials: The role of the c-statistic. *BMC Med Res Methodol*. 2016;16:9.
- 181. Stuart EA, Rubin DB. Best practices in quasi-experimental designs: Matching methods for causal inference. In: Osborne JW, ed. *Best Practices in Quantitative Methods*. Thousand Oaks, CA: Sage; 2007:155-176
- 182. Austin PC, Stuart EA. Moving towards best practice when using inverse probability of treatment weighting (IPTW) using the propensity score to estimate causal treatment effects in observational studies. *Stat Med.* 2015;34(28):3661-3679.
- 183. Taft AJ, Small R, Hegarty KL, Watson LF, Gold L, Lumley JA. Mothers' AdvocateS In the Community (MOSAIC)--Non-professional mentor support to reduce intimate partner violence and depression in mothers: A cluster randomised trial in primary care. *BMC Public Health*. 2011;11:178.
- 184. Vickers AJ, Altman DG. Statistics notes: Analysing controlled trials with baseline and follow up measurements. *BMJ*. 2001;323(7321):1123-1124.
- 185. Wolfinger R, O'Connell M. Generalized linear mixed models: A pseudo-likelihood approach. *J Stat Comput Simul*. 1993;48:233-243.
- 186. Pinheiro JC, Bates DM. Approximations to the log-likelihood function in the nonlinear mixed-effects model. *J Comput Graph Statist*. 1995;4(12-35).
- 187. Murray DM. Statistical models appropriate for designs often used in group-randomized trials. *Stat Med.* 2001;20:1373-1385.
- 188. Pham H. Springer Handbook of Engineering Statistics. New York, NY: Springer; 2006.
- 189. Fleiss JL. Some thoughts on two-sided tests. J Controlled Clin Trials. 1987;8:394.
- 190. Viswanathan M, Eng E, Ammerman A,... Rhodes SD, et al. *Community-based participatory research: Assessing the evidence*. Rockville, MD: Agency for Healthcare Research and Quality; July 2004. 99.
- 191. Hergenrather KC, Rhodes SD. Community-based participatory research: Applications for research in health and disability. In: Knoll T, ed. *Focus on Disability: Trends in Research and Application*. Vol 2. New York: NY: Nova Science; 2008:59-87.

- 192. Israel BA, Eng E, Schulz AJ, Parker EA. Introduction to methods in community-based participatory research for health. In: Israel BA, Eng E, Schulz AJ, Parker EA, eds. *Methods in Community-Based Participatory Research*. San Francisco, CA: Jossey-Bass; 2005.
- 193. Baquero B, Goldman SN, Simán F, Muqueeth S, Eng E, Rhodes SD. Mi Cuerpo, Nuestro Responsabilidad: Using Photovoice to describe the assets and barriers to reproductive health among Latinas. *J Health Dispar Res Pract.* 2014;7(1):65-83.
- 194. Freire P. Pedagogy of the Oppressed. New York, NY: Herder and Herder; 1970.
- 195. Wallerstein N. Empowerment education applied to youth. In: Matiella AC, ed. *The Multicultural Challenge in Health Education*. Santa Cruz, CA: ETR Associates; 1994:153-176.
- 196. Becker AB, Israel BA, Gustat J, Reyes AG, Allen AJ. Strategies and techniques for effective group process in CBPR partnerships. In: Israel BA, Eng E, Schulz AJ, Parker EA, eds. *Methods in Community-Based Participatory Research for Health*. San Francisco, CA: Jossey-Bass; 2013:69-95.
- 197. Green LW, Krueter M, Krueter MW. *Health Promotion Planning: An Educational and Environmental Approach.* 3 ed. Mountain View, CA: Mayfield Publications; 1999.
- 198. Green LW, O'Neill M, Westphal M, Morisky D. The challenges of participatory action research for health promotion. *Promot Educ.* 1996;3(4):3-5.
- 199. Eng E, Strazza K, Rhodes SD, et al. Insiders and outsiders assess who is "the community":
- Participant observation, key informant interview, focus group interview, and community forum. In: Israel BA, Eng E, Schulz AJ, Parker E, eds. *Methods for Conducting Community-Based Participatory Research for Health*. 2 ed. San Francisco, CA: Jossey-Bass; 2013:133-160.
- 200. Krogstad JM. *Hispanics Have Accounted for More Than Half of Total U.S. Population Growth Since 2010.* Washington, DC: Pew Research Center. 2020.
- 201. Streiner DL, Norman GR. *Health Measurement Scales: A Practical Guide to their Development and Use.* Oxford: Oxford University Press; 1995.